CLINICAL TRIAL: NCT05255276
Title: A Phase 1 Open-label, Two-cohort, One-sequence Crossover Study to Investigator the Effect of P-glycoprotien Inhibitor (Itraconazole) and Inducer (Rifampin) on the Pharmacokinetics, Safety, and Tolerability of Sitravatinib in Health Subjects
Brief Title: PK Study to Assess Drug-drug Interaction Between Sitravatinib and a P-gp Inducer and an Inhibitor.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 516-013
Record Dates: First submitted 2022-02-10; First posted 2022-02-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adults
MeSH Terms: interventions — sitravatinib; Itraconazole; Pantoprazole; Rifampin; Famotidine

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, single-center, open-label, 2-cohort, 1-sequence crossover study to investigate the effect of coadministration of a P glycoprotein (P-gp) inhibitor, itraconazole, (Cohort 1) and a P-gp inducer, rifampin, (Cohort 2) in healthy subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Treatment A (Active Comparator): A single-dose administration of sitravatinib malate 50 mg on Day 1. Day 12, a single dose of sitravatinib malate 50 mg will be will be followed by a 72-hour PK sample collection period. Subjects will be discharged from the CRU on Day 4 after collection of 72-hour postdose PK sample and completion of all required study procedures.
  Interventions: Drug: Sitravatinib 50 mg
- Group 1 Treatment B (Active Comparator): On Days 9 to 11, itraconazole 200 mg will be administered QD in the morning. On Day 12, a single dose of sitravatinib malate 50 mg will be coadministered with itraconazole. Itraconazole QD dosing will continue on Days 13 to 18 to maintain steady state during the PK sample collection period.
  Interventions: Drug: Itraconazole
- Group 2 Treatment A (Active Comparator): A single-dose administration of sitravatinib malate 100 mg on Day 1 will be followed by a 72-hour PK sample collection period. Subjects will be discharged from the CRU on Day 4 after collection of 72-hour postdose PK sample and completion of all required study procedures.
  Interventions: Drug: Sitravatinib 100 mg
- Group 2 Treatment B (Active Comparator): On Days 9 to 15, rifampin 600 mg will be administered QD in the morning. On Day 16, a single dose of sitravatinib malate 100 mg will be coadministered with rifampin followed by a 72 hour PK sample collection period. Rifampin QD dosing will continue on Days 17 to 22 to maintain steady state during the PK sample collection period.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Sitravatinib 50 mg — 50 mg Sitravatinib on Day 1 (Group 1A)
  Other Names: MGCD516
  Arms: Group 1 Treatment A
Drug: Sitravatinib 100 mg — 100 mg Sitravatinib on Day 1 (Group 2A)
  Other Names: MGCD516
  Arms: Group 2 Treatment A
Drug: Itraconazole — Itraconazole QD from Day 9 to Day 18, and Sitravatinib 50 mg at Day 12 (Group 1B)
  Other Names: Protonix
  Arms: Group 1 Treatment B
Drug: Rifampin — Rifampin QD from Day 9 to Day 22, and Sitravatinib 100 mg at Day 16 (Group 2B)
  Other Names: Pepcid
  Arms: Group 2 Treatment B

SUMMARY:
A Phase 1 Open-label, Two-cohort, One-sequence Crossover Study to Investigate the Effect of P glycoprotein Inhibitor (Itraconazole) and Inducer (Rifampin) on the Pharmacokinetics, Safety, and Tolerability of Sitravatinib in Healthy Subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and/or check-in, as assessed by the investigator (or qualified designee).
* Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at screening and check-in. Females of childbearing potential must agree to use contraception.
* Male subjects must agree to use contraception.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Key Exclusion Criteria:

* Significant history of clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, any components of the IMP, or other substance (not including seasonal allergies), unless approved by the investigator.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications. (Uncomplicated appendectomy and hernia repair are allowed. Cholecystectomy is not allowed.)
* History of Gilbert's syndrome or suspicion of Gilbert's syndrome based on elevated total and indirect bilirubin (may be confirmed by repeat).
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to study drug administration on Day 1 of Period 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax (sitravatinib) | Up to Day 168 hours after dosing
  Maximum observed plasma concentration
Pharmacokinetics - AUC∞ (sitravatinib) | Up to 168 hours after dosing
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUClast (sitravatinib) | Up to 168 hours after dosing
  Area under the curve from time zero to the last measured time point
Pharmacokinetics - tmax (sitravatinib) | Up to 168 hours after dosing
  Terminal elimination half-life
Pharmacokinetics - CL/F (sitravatinib) | Up to 168 hours after dosing
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - Vz/F (sitravatinib) | Up to 168 hours after dosing
  Apparent volume of distribution when dosed orally
Pharmacokinetics - uf (sitravatinib) | Up to 168 hours after dosing
  Unbound fraction

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 12 weeks from screening
  Incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Drug Development Clinical Research Unit, Dallas, Texas, United States